CLINICAL TRIAL: NCT01717287
Title: A Phase II, Multicenter, Open-Label, Noncomparative Study of Raltegravir (MK-0518) in Two Oral Formulations in Combination With Other Antiretroviral Agents to Evaluate the Safety, Tolerability, and Antiretroviral Activity in HIV-1 Infected Russian Children and Adolescents
Brief Title: A Study of the Safety, Tolerability, and Antiretroviral Activity of Raltegravir (MK-0518) in Combination With Other Antiretroviral Therapies in Russian Children and Adolescents Infected With Human Immunodeficiency Virus (HIV-1) (MK-0518-248)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0518-248
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Results first posted 2014-07-29 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltegravir Film-coated Tablet (Experimental): Raltegravir film-coated tablet 400 mg administered orally twice-daily, in combination with other anti-retroviral therapy for 24 weeks
  Interventions: Drug: Raltegravir Film-coated Tablet; Drug: Other Anti-Retroviral Therapy
- Raltegravir Chewable Tablet (Experimental): Raltegravir chewable tablet weight-based dose up to 300 mg administered orally twice-daily, in combination with other anti-retroviral therapy for 24 weeks
  Interventions: Drug: Raltegravir Chewable Tablet; Drug: Other Anti-Retroviral Therapy

INTERVENTIONS:
Drug: Raltegravir Film-coated Tablet
  Other Names: ISENTRESS®; MK-0518
  Arms: Raltegravir Film-coated Tablet
Drug: Raltegravir Chewable Tablet
  Other Names: ISENTRESS®; MK-0518
  Arms: Raltegravir Chewable Tablet
Drug: Other Anti-Retroviral Therapy — At baseline, the investigator selected the other anti-retroviral therapies to be used in combination with raltegravir based on current treatment guidelines, the participant's treatment history, and prior anti-retroviral resistance testing

SUMMARY:
This multicenter, open-label, noncomparative study evaluates two oral formulations of raltegravir (MK-0518, film-coated tablet and chewable tablet) in combination with other antiretroviral agents for safety, tolerability, and antiretroviral activity in treatment-naive or treatment-experienced Russian children and adolescents infected with human immunodeficiency virus-1 (HIV-1).

As raltegravir is indicated in combination with other antiretroviral therapies (ARTs) for the treatment of HIV-1 infection in pediatric patients in the United States (US), this study is designed to gain local treatment experience on the use

of raltegravir in the pediatric HIV-infected population in Russia.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Weight of at least 7 kg
* HIV RNA ≥1000 copies/mL within 45 days before study treatment
* Participants of reproductive potential and sexually active agree to remain

abstinent or use (or have their partner use) an acceptable method of birth control throughout the study.

Exclusion Criteria:

* Females pregnant or breast-feeding, or expecting to conceive or donate eggs

during the study; males planning to impregnate or provide sperm donation

during the study

* Use of any non-antiretroviral (ART) investigational agents within one month before study treatment
* Current (active) diagnosis of acute hepatitis or chronic hepatitis other than stable chronic Hepatitis B and/or C
* Prior or current use of raltegravir
* Use of another experimental HIV-integrase inhibitor
* History or current evidence of any condition, therapy, laboratory

abnormality, or other circumstance that might confound the results of the study, or interfere with participation for the full duration of the study

* Requires or is anticipated to require any prohibited medications
* Use of immunosuppressive therapy within 30 days before beginning

raltegravir study treatment; short courses of corticosteroids are permitted.

* History of malignancy
* Current treatment for active tuberculosis infection
* Use of recreational or illicit drugs or a recent history (within the

last year) of drug or alcohol abuse or dependence

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-11-16 (Actual); Primary Completion 2013-12-11 (Actual); Study Completion 2013-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0518-248&kw=0518-248&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Film-coated tablets were administered to participants >=12 years old and to those 6 to <12 years old who weighed >=25 kg and could swallow pills. A weight-based dose of chewable tablets was administered to participants 6 to <12 years old who could not swallow pills or preferred the chewable formulation, and to participants 2 to <6 years old
Period: Overall Study
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Started | 4 | 28
Completed | 4 | 25
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet | Total
Number analyzed (Participants) | 4 | 28 | 32
Age, Customized [Number; unit: Participants]
  2 to <6 years | 0 | 11 | 11
  6 to <12 years | 2 | 17 | 19
  12 to <18 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 16 | 17
  Male | 3 | 12 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Clinical Adverse Experience
Description: A clinical adverse experience is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study drug is also an adverse experience.
Time Frame: Up to Week 26
Population: All patients as treated population included all enrolled participants who received at least one dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Number analyzed (Participants) | 4 | 28
Percentage of participants | 0.0 | 42.9

2. Primary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to a Clinical Adverse Experience
Description: as for outcome 1
Time Frame: Up to Week 24
Population: All patients as treated population included all enrolled participants who received at least one dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Number analyzed (Participants) | 4 | 28
Percentage of participants | 0.0 | 0.0

3. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4) Cell Count
Description: This outcome is a measure of immunological response to treatment
Time Frame: Baseline and Week 24
Population: The population analyzed included all participants who received at least one dose of study drug, had baseline evaluation (required for change from baseline endpoints only), and had Week 24 evaluation
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Number analyzed (Participants) | 3 | 24
cells/mm^3 | 30.3 [-178.6 to 239.2] | 296.3 [133.6 to 458.9]

4. Secondary Outcome: Change From Baseline in CD4 Cell Percentage
Description: This outcome is a measure of immunological response to treatment
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Number analyzed (Participants) | 3 | 24
Percentage change | 4.0 [-5.0 to 13.0] | 6.0 [3.8 to 8.1]

5. Primary Outcome: Percentage of Participants With at Least One Laboratory Adverse Experience
Description: A laboratory adverse experience is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study drug is also an adverse experience.
Time Frame: Up to Week 26
Population: All patients as treated population included all enrolled participants who received at least one dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Number analyzed (Participants) | 4 | 28
Percentage of participants | 0.0 | 3.6

6. Primary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to a Laboratory Adverse Experience
Description: as for outcome 5
Time Frame: Up to Week 24
Population: All patients as treated population included all enrolled participants who received at least one dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Number analyzed (Participants) | 4 | 28
Percentage of participants | 0.0 | 0.0

7. Secondary Outcome: Percentage of Participants Achieving >=1 log10 Reduction From Baseline in Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) or Had an HIV RNA Assessment of <200 Copies/mL
Description: This outcome is a measure of virological (anti-retroviral) response to treatment. Plasma HIV RNA was measured using the Abbott RealTime HIV-1 assay, which has a linear range of 40 HIV RNA copies/mL to 10 million HIV RNA copies/mL
Time Frame: Week 24
Population: Full analysis set included all participants who received at least one dose of study drug, had baseline evaluation (required for change from baseline endpoints only), and had at least one postbaseline evaluation
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Number analyzed (Participants) | 4 | 25
Percentage of participants | 75.0 [19.4 to 99.4] | 88.0 [68.8 to 97.5]

8. Secondary Outcome: Percentage of Participants Achieving HIV RNA <40 Copies/mL
Description: as for outcome 7
Time Frame: Week 24
Population: Full analysis set included all participants who received at least one dose of study drug, had baseline evaluation, and had at least one postbaseline evaluation
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Number analyzed (Participants) | 4 | 25
Percentage of participants | 50.0 [6.8 to 93.2] | 44.0 [24.4 to 65.1]

9. Secondary Outcome: Percentage of Participants Achieving HIV RNA <200 Copies/mL
Description: as for outcome 7
Time Frame: Week 24
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Number analyzed (Participants) | 4 | 25
Percentage of participants | 50.0 [6.8 to 93.2] | 76.0 [54.9 to 90.6]

ADVERSE EVENTS:
Time Frame: Up to Week 26
Arm/Group | Raltegravir Film-coated Tablet | Raltegravir Chewable Tablet
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/28
Other Adverse Events (participants affected / at risk) | 0/4 | 8/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir Film-coated Tablet (N=4) | Raltegravir Chewable Tablet (N=28)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (6)
Otitis media (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.